CLINICAL TRIAL: NCT07098377
Title: Gut, Nasopharyngeal, and Skin Microbiota in Children With Severe Burn Injury: the Role in Infectious Complications in Burn Injury
Brief Title: Microbiota in Children With Severe Burn Injury
Acronym: MIBUS
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7327
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-03

CONDITIONS: Burn
Keywords: burns; microbiota; sepsis
MeSH Terms: conditions — Burns; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- burns affected
  Interventions: Diagnostic Test: nasopharyngeal swab for biological sample analysis

INTERVENTIONS:
Diagnostic Test: nasopharyngeal swab for biological sample analysis — nasopharyngeal swab for biological sample analysis

SUMMARY:
The research protocol consists of taking aliquots of biological specimens from skin swabs, nasopharyngeal swabs, and fecal swabs. the samples will be taken at time 0 of admission to the Pediatric ICU, one week after admission, and two weeks after admission to compare the bacterial populations present at the different sampling sites.

DETAILED DESCRIPTION:
Pediatric burns (0-14 years) make up 26% of emergency room admissions for burns, with 73% of cases in children under 5 years old. The most common burns are thermal from boiling liquids, followed by open flames and fireworks. Severe burns (>20% of body surface area) provoke a systemic inflammatory response that causes hypovolemia, tissue hypoperfusion, and metabolic stress, establishing a vicious cycle that is difficult to break.

Burn trauma can also compromise the intestinal barrier, composed of cellular junctions (tight junctions), damage to which increases intestinal permeability. This promotes the passage of luminal contents into the systemic circulation, aggravating the immune and inflammatory response. Gut dysfunction is often accompanied by dysbiosis of the microbiota, with risk of bacterial translocation to sterile organs (liver, lungs, brain), contributing to systemic complications in critically ill patients.

The study hypothesizes that burn trauma increases intestinal permeability, promoting bacterial translocation and anticipating infectious complications. Analyzing microbial populations at exposed sites (skin, gut, BAL) during trauma and pediatric ICU care may help to better understand the origin of septic complications.

ELIGIBILITY:
Inclusion Criteria:

* signs and/or symptoms of burn injury

Exclusion Criteria:

* major congenital malformation
* Antibiotic treatment 48 hours prior to admission
* failure to provide informed consent to participate in the protocol

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children suffering from burn trauma with signs and symptoms of burns, without antibiotic therapy in the previous 48 hours and without major congenital malformations. Authorization for data processing and participation in the study by the patient or their legal guardians is also considered.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
intestinal microbiota variation in burnt children | 21 days
  concentration of microbiota population in pediatric population severely burnt

CONTACTS AND LOCATIONS:
Overall Officials: Orazio Genovese, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
results microbiota variation in severely burnt children
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: two years